CLINICAL TRIAL: NCT04633785
Title: Validation of Wrist Type Oscillometric Blood Pressure Monitorings
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-11-001CC
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Blood Pressure
Keywords: oscillometric; wrist blood pressure monitor; sphygmomanometer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- wrist BP
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There are no interventions in this study. The mercury sphygmomanometer and the wrist sphygmomanometer will be used in this study to collect blood pressure values from the study subjects.

SUMMARY:
Since the wrist devices have the advantage of being smaller, lighter, and more inexpensive than the upper arm devices, wrist devices become increasingly popular. However, it is of utmost importance to ensure that the BP measuring device can measure BP accurately. This study will be aimed to validate a wrist type oscillometric blood pressure monitoring with reference to the brachial blood pressure measured by auscultatory method with a mercury sphygmomanometer.

DETAILED DESCRIPTION:
High blood pressure (BP) is one of the major cardiovascular risk factors in adults. Home blood pressure monitoring is superior to office-based measurements for prediction of the future development of cardiovascular diseases and is recommended by major guidelines. To monitor BP at home, patients can use devices that measure BP either at the arm or at the wrist.

Among BP monitors, the wrist device is relatively easy to use, as the cuff can be used with one hand easily and correctly around the wrist than around the arm, and undressing is not necessary. Since the wrist devices have the advantage of being smaller, lighter, and more inexpensive than the upper arm devices, wrist devices become increasingly popular. However, it is of utmost importance to ensure that the BP measuring device can measure BP accurately. To make sure the performance of these devices, several guidelines have proposed protocols to validate these devices. This study will be aimed to validate a wrist type oscillometric blood pressure monitoring with reference to the brachial blood pressure measured by auscultatory method with a mercury sphygmomanometer.

ELIGIBILITY:
Inclusion Criteria:

* above 12 years old

Exclusion Criteria:

* unclear Korotkoff sounds
* wrist circumference outside of the designated range (13.5-23 cm)
* arrhythmias

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from outpatient clinics at Taipei Veterans General Hospital from 2020 to 2021. A total of 100 subjects will be enrolled in the study, and informed consent forms will be obtained from before measurements. In accordance with the ANSI/AAMI/ISO, subjects will be screened to ensure that sex, age, wrist circumference, and BP readings fulfilled the participation requirements described in those protocols. If subjects aged less than 12 years old, having wrist circumference outside of the designated range (13.5-23 cm), having arrhythmias, who moved their arms or bodies during the BP measurements, and have unclear Korotkoff sounds will be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Validation | 7 months
  The present study will be aimed to evaluate the accuracy of the wrist type oscillometric blood pressure monitorings.

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Min Cheng, M.D., Ph.D., Study Director — Center for Evidence-based Medicine, Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: No